CLINICAL TRIAL: NCT00630110
Title: Study of the Vascular Disrupting Agent NPI-2358 in Combination With Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Phase 1/2 Study of Vascular Disrupting Agent NPI-2358 + Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nereus Pharmaceuticals, Inc. (Industry)
Responsible Party: Kristine C. Federico, RN BSN - Director Clinical Development, Nereus Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPI-2358-101
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Cancer
Keywords: Non Small Cell Lung
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel; NPI 2358

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- docetaxel (Active Comparator): docetaxel (75 mg/m2)
  Interventions: Drug: docetaxel
- NPI-2358 + docetaxel (Experimental): NPI-2358 (30 mg/m2) + docetaxel (75 mg/m2)
  Interventions: Drug: NPI-2358 + docetaxel

INTERVENTIONS:
Drug: docetaxel — docetaxel (75 mg/m2)
  Other Names: docetaxel (Taxotere)
  Arms: docetaxel
Drug: NPI-2358 + docetaxel — NPI-2358 (30 mg/m2) + docetaxel (75 mg/m2)
  Other Names: NPI-2358; docetaxel (Taxotere)
  Arms: NPI-2358 + docetaxel

SUMMARY:
This is a clinical trial examining the vascular disrupting agent NPI-2358 combined with docetaxel in patients with advanced non-small cell lung cancer (NSCLC). The formation of new blood vessels (angiogenesis) is an important component of tumor growth, vascular disrupting agents are intended to target the differences between these tumor blood vessels and the blood vessels in normal tissues.

DETAILED DESCRIPTION:
This is a clinical trial examining the vascular disrupting agent NPI-2358 combined with docetaxel in patients with advanced non-small cell lung cancer (NSCLC). The formation of new blood vessels (angiogenesis) is an important component of tumor growth, vascular disrupting agents are intended to target the differences between these tumor blood vessels and the blood vessels in normal tissues. There are indications of advantages in combining vascular disrupting agents with standard agents in the treatment of advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Male and females ≥ 18 years of age
* ECOG performance status ≤ 1
* Pathologically or histologically confirmed advanced non-small cell lung cancer (unresectable Stage IIIb or IV) that has progressed after treatment with at least one chemotherapy regimen; measurable disease is not required for enrollment into this trial
* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to Grade ≤ 2
* Signed informed consent

Exclusion Criteria:

* Administration of certain chemotherapy, biological, immunotherapy, radiation therapy, surgery or investigational agent within specified time frames
* Significant cardiac history
* Prior treatment with tumor vascular disruptive agents
* Seizure disorder
* Brain metastases
* Active uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy
* Known infection with human immunodeficiency virus (HIV), or active hepatitis A, B, or C
* Patients with a prior hypersensitivity reaction to product components
* Pregnant or breast-feeding women.
* Concurrent, active second malignancy for which the patient is receiving therapy, excluding basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Unwilling or unable to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Compare overall survival of patients treated with docetaxel to patients treated with docetaxel + NPI-2358 | Continuous

SECONDARY OUTCOMES:
Compare response rate, duration of response, 6-month survival, progression free survival and safety. | Continuous
Pharmacokinetics | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Spear, MD, Study Director — Chief Medical Officer, Nereus Pharmaceuticals, Inc
Locations (36):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - San Diego Pacific Oncology & Hematology Associates, Encinitas, California
  - University San Diego Moores Cancer Center, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Premiere Oncology, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University Texas Health Science Center at San Antonio (CTRC), San Antonio, Texas
- Argentina (6):
  - Policlinica Privada Instituto de Medicina Nuclear, Bahía Blanca
  - Hospital Britanico, Capital Federal
  - Instituto Oncologico De Cordoba, Córdoba
  - Clinica Universitaria Privada Reina Fabiola, Córdoba
  - Caici Centro de Asistencia e Investigacion Clinica Integral, Rosario
  - Hospital del Centrenario, Rosario
- Australia (3):
  - Mater Adult Hospital, South Brisbane, Queensland
  - Bendigo Health Care Group, Bendigo, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (8):
  - Fundacap Pip XII Hospital do Cancer de Barretos, Barretos
  - Hospital Erasto Gaertner Liga do Combate as Cancer, Curitiba
  - Associacao Hospital de Caridade Ijui, Ijuí
  - Hospital Sao Lucas, Porte Alegre
  - Hospital de clinicas de Porto Alegre, Porto Alegre
  - Clinionco-Clinica de Oncologia de Porto Alegre, Porto Alegre
  - Hosp.das Clinicas da Univ.de Sao Paulo, São Paulo
  - Instituto do Cancer Aenaldo Vieira de Carvahlo, São Paulo
- Chile (2):
  - Instituto Nacional del Cancer Oncology, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- India (9):
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Apollo Speciality Hospital, Chennai
  - Apollo Hospital, Hyderabad
  - SEAROC Cancer Centre S.K. Soni Hospital, Jaipur
  - Subodh Mitra Cancer Hospital & Research Centre, Kolkata
  - Tata Memorial Hospital, Mumbai
  - Ruby Hall Clinic, Pune
  - Andhra Medical College, Visakhapatnam